CLINICAL TRIAL: NCT03929575
Title: Effects of Herbal Supplements on Endurance Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Principal Investigator, Todd Hagobian, Principal Investigator, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: CPKINE454
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Exercise Performance

STUDY DESIGN:
Intervention Model Description: Blocked-randomized, crossover design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo of calcium (Placebo Comparator): Participants will consume 250 mg of calcium
  Interventions: Dietary Supplement: Placebo of calcium
- Rhodiola (Experimental): Participants will consume 250 mg of Rhodiola
  Interventions: Dietary Supplement: Rhodiola
- Rhodiola and Cordyceps (Experimental): Participants will consume a combination of 250 mg of Rhodiola and 225 mg of Cordyceps
  Interventions: Dietary Supplement: Rhodiola and Cordyceps

INTERVENTIONS:
Dietary Supplement: Placebo of calcium — Ingestion of 250 mg of calcium
  Arms: Placebo of calcium
Dietary Supplement: Rhodiola — Ingestion of 250 mg of Rhodiola
  Arms: Rhodiola
Dietary Supplement: Rhodiola and Cordyceps — Ingestion of 250 mg of Rhodiola and 225 mg of Cordyceps
  Arms: Rhodiola and Cordyceps

SUMMARY:
Cordyceps and Rhodiola are two common herbal supplements marketed and consumed as adaptogens to athletes with regard to enhanced performance. The effects of these supplements has been well studied in animals but whether or not the same effects translate to humans is still unclear. Thus, the primary purpose of this study is to determine whether combined supplementation of Rhodiola and Cordyceps, compared to Rhodiola alone and placebo, will demonstrate a greater improvement in oxygen consumption (ie. VO2 max).

DETAILED DESCRIPTION:
Herbal supplements are consumed worldwide with surveys approximating five billion dollars spent annually by consumers in the United States alone. Herbal supplements, such as Rhodiola and Cordyceps, both of which are considered to be adaptogens, remain popular among athletes. These adaptogens act as antioxidants, which have been speculated to confer endurance performance benefits by delaying muscle fatigue via the attenuation of muscle damage accumulation and its related by-products during prolonged or exhaustive exercise. Nevertheless, previous research investigating the individual effects of Rhodiola and Cordyceps on aerobic training performance remain equivocal. Moreover, literature elucidating the potential additive effects of Rhodiola and Cordyceps in human subjects are scarce. Therefore, the purpose of the present study is to determine the acute, additive influence of oral Rhodiola and Cordyceps supplementation on VO2 max, with secondary variables of interest being plasma glucose and lactate concentration, and measures of gastrointestinal distress.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 18.5 and 35 kg/m^2
* Non-smoking (assessed by Health History Questionnaire)
* English-speaking
* Regular participation in physical activity (>4 hours per week)

Exclusion Criteria:

* Medical conditions that prohibit physical activity (assessed by Health History Questionnaire)
* Pregnant women or women expecting/trying to become pregnant
* BMI greater than or equal to 35 kg/m^2
* Current smoker (assessed by Health History Questionnaire)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
VO2 max | 90 minutes after baseline
  Maximum oxygen consumption using the Bruce Protocol

SECONDARY OUTCOMES:
Gastrointestinal symptoms questionnaire | Baseline, 90 minutes, 110 minutes
  Section 1 contains 6 questions assessing upper abdominal problems (reflux, heartburn, bloating, cramps, vomiting, and nausea). Section 2 contains 7 questions assessing lower abdominal problems (intestinal cramps, flatulence, urge to defecate, left abdominal pain, right abdominal pain, loose stool, and diarrhea). Section 3 contains 4 questions assessing systematic problems (dizziness, headache, muscle cramp, and urge to urinate). Each of the 17 questions is answered using a 10-point scale ranging from 0 (no problem at all) to 10 (the worst it has ever been). Each of the 3 sections will be scored separately. Section 1 will be scored on a scale of 0-60. Section 2 will be scored on a scale of 0-70. Section 3 will be scored on a scale of 0-40.
Blood glucose | Baseline, 90 minutes, 110 minutes
  Plasma glucose assessed by finger stick
Blood lactate | Baseline, 90 minutes, 110 minutes
  Plasma lactate assessed by finger stick

CONTACTS AND LOCATIONS:
Overall Officials: Todd Hagobian, PhD, Principal Investigator — California Polytechnic State University-San Luis Obispo
Locations (1):
- California Polytechnic State University, San Luis Obispo, California, United States

IPD SHARING:
Plan to Share IPD: No